CLINICAL TRIAL: NCT03379142
Title: Faith Based Pilot Intervention to Reduce Tobacco Use Among Somali Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FMCH-2017-25736
Record Dates: First submitted 2017-11-29; First posted 2017-12-20 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Tobacco Use; Faith-Based; Community-engaged; Text Messaging
Keywords: Faith-Based; Community-engaged; Text messaging; Tobacco
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioral: Faith-Based messages (Other): We will send faith-based messages one week prior to Ramadan and twice a day during Ramadan.
  Interventions: Behavioral: Faith-Based messages

INTERVENTIONS:
Behavioral: Faith-Based messages — We will send out faith based text messages on a weekly basis for the one week prior to the start of Ramadan, then twice a day during the Ramadan period that will encourage smoking cessation and continue to encourage change of behavior. The faith-based messages will be incorporated with messages drawn from the Smokefree.gov Mobile Interventions QuitNowTXT Message Library. These messages will be geared towards reminding the smokers that as Ramadan is coming closer they need to consider the effects that smoking may have on their health and should consider taking steps towards quitting.

SUMMARY:
1.1 In the last five years, representatives of WellShare International and the University of Minnesota have engaged a large community of Muslims of Somali descent in the Twin Cities of Minnesota in a community-academic research program to understand smoking and cessation behaviors. This followed research by WellShare International which discovered a smoking prevalence among Somali men of 44%, which is nearly three times that of the general population (14.4%) in Minnesota. More recently, pilot data from ecological momentary assessments (EMA) conducted by WellShare International and the University of Minnesota Program in Health Disparities Research before and during Ramadan, showed that the majority of smokers achieved spontaneous significant reductions in cigarettes smoked per day during Ramadan. Guided by the NIH Stage Based Intervention Development Model, this study aims to understand the processes underlying smoking reduction and cessation during Ramadan. The investigators plan to harness this knowledge and develop a culturally-tailored, faith-based smoking cessation intervention (Stage 1). The investigators also plan to assess the feasibility of the new culturally-tailored smoking cessation intervention by conducting a pilot study (Stage 2).

The study aims are as follows:

Aim 1: To develop a faith-based, community-informed innovative smoking cessation intervention for use with a Somali immigrant population in Minnesota:

Aim 2: To assess the feasibility of a faith-based smoking cessation intervention delivered via a mobile phone during the Ramadan period:

This pilot study will test a protocol for use of faith based text messages, as informed by the scholarly work of the Imams, Community Advisory Group (CAG) and focus groups conducted in Stage 1.

DETAILED DESCRIPTION:
Smoking Prevalence in the Muslim communities: Although significant declines in cigarette smoking prevalence have been realized in the United States (U.S.), this decline is not universal. Muslim communities continue to have disproportionately high smoking prevalence rates. For example, one of WellShare International's studies showed a smoking prevalence rate of 44.1% among Somali adult (predominantly Muslim) men in Minnesota, compared to the average smoking rate for adult men in Minnesota (14.4%) and in the United States of 17.8%. Despite ample evidence that pharmacotherapy and counselling are effective for smoking cessation in the general population, no one has identified effective ways to extend these benefits to the Muslim communities and the U.S.'s largest Somali population which resides in Minnesota. Even when readily available, such aids seem to be underutilized, reflecting the commonly held belief among Muslims that giving up smoking primarily requires only will power. Although approaches that draw on the need for will power around the Ramadan fast (during which smoking is prohibited during daylight hours) have been considered, no systematic attempt has been made to make effective evidence-based smoking cessation methods available leveraged on the Ramadan. Muslim smokers face yet another challenge during the holy month of Ramadan, where adherence to medications during this month has been documented as challenging. However, because cigarette smoking continues to be the leading cause of morbidity and mortality, it is critical to identify evidence-based methods for promoting adherence to known effective methods for reducing tobacco related health disparities in this underserved minority population in Minnesota.

ELIGIBILITY:
Inclusion Criteria:

* Somali Male
* 18 years of age or older
* Can read either Somali or English (Non English Speaking Participants will be included)
* Current smokers defined as smoking ≥ 1 cigarette per day
* Self-report of smoking ≥ 100 cigarettes in their lifetime
* Willingness to use nicotine patch or other selected pharmacotherapy
* Possess a working mobile phone with texting
* Planning to fast during Ramadan

Exclusion Criteria:

* Currently using any form of smoking cessation service
* Any medical contraindication
* Current history or in past 6 months of a psychotic disorder
* Suicidal ideation
* Cognitive impairment
* Any other medical condition that, in the opinion of the investigator, may interfere with the patient's ability to successfully and safely complete the study

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Somali Male smokers
Enrollment: 50 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Participants Adherence to the Intervention | 8 weeks
  Real time smoking cravings and urges, as well as the number of cigarettes smoked in each time period, will be measured via ecological momentary assessment (EMA) in a sample of Muslim male smokers who are fasting during Ramadan. Participants will be enrolled in this study if they are current smokers and are going to fast throughout Ramadan. Analyses will use data collected via a RedCap survey at random time points (3 times per day, 2 times a week) during Ramadan. In the analysis, 4 time blocks (pre sunrise [4:30am-9:00am], day time [9:01am-3:00pm], pre sunset [3:01pm-9:00pm] and breaking fast [9:01pm-4:29am]) will be used for analysis.

SECONDARY OUTCOMES:
smoking cessation | 8 weeks
  CO breath test at week 4 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Olamide Ojo-Fati, MD MPH, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - WellShare International, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pratt R, Ojo-Fati O, DuBois D, Okuyemi K, Graham AL, Mohamed S, Janowiec M, Kahin A, Mahamud A, Tessier KM, Busch AM, Joseph AM. Testing the Feasibility and Acceptability of a Religiously-Tailored Text Messaging Intervention to Reduce Smoking Among Somali Muslim Men During Ramadan. Nicotine Tob Res. 2021 Aug 4;23(8):1283-1290. doi: 10.1093/ntr/ntaa260. PMID 33277991